CLINICAL TRIAL: NCT07136038
Title: Prevention and Education for RED-S Through Fueling Outcomes and Research in Metabolic Health
Brief Title: Preventing Athlete Under-fueling Through Nutrition.
Acronym: PERFORM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY20250865
Record Dates: First submitted 2025-08-18; First posted 2025-08-22 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Athlete; Relative Energy Deficiency in Sport; Low Energy Availability
Keywords: collegiate; sport; lean body mass; fat mass
MeSH Terms: conditions — Relative Energy Deficiency in Sport | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Single-group, open label nutrition intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Athletes (Experimental)
  Interventions: Behavioral: Low Energy Availability Screening and Nutrition Support

INTERVENTIONS:
Behavioral: Low Energy Availability Screening and Nutrition Support — Athletes will receive screening for low energy availability, strength and body composition assessments and receive nutrition support from a sports dietitian over the competitive season.

SUMMARY:
The goal is to improve nutrition screening and support for Division III athletes.

The study will use standard, low-risk nutrition screening methods, such as measuring height, weight, grip strength, and body composition, as well as having athletes complete questionnaires. Dietitians trained in sports nutrition will provide nutrition advice based on these screenings.

Data will be collected at three points during the season: before the season starts, mid-season, and after the season ends. This study builds on earlier research conducted at Case Western Reserve University that showed nutrition support can improve athletes' health and performance.

DETAILED DESCRIPTION:
OBJECTIVES: Combat student athletes' under fueling before, during and after the competitive season and assess financial feasibility for scaling to the university level.

STUDY OVERVIEW: This project proposes an open label, pilot research endeavor between the Department of Nutrition at Case Western Reserve University (CWRU), Pennington Biomedical Research Center (PBRC) and the NCAA Division III CWRU Athletic Department. The proposed study design will implement improved nutrition screening and support, applying standard-of-practice processes that are used at the highest level of collegiate sport (Division I) modified for the Division III athlete. This study will utilize minimal-risk/standard-of-care nutrition screening procedures along with standard-of-care nutrition advice from dietitians trained in sports nutrition. All athletes will be screened with minimal risk items such as anthropometrics, questionnaires, grip strength and body composition testing. While additional voluntary metrics will be provided in a subset of individuals based on team and individual availability and include aerobic fitness (VO2), resting metabolic rate, physical activity, body composition and sports performance. Data will be collected at three timepoints: pre-season, mid-season, and post-season. Notably, this work expands upon the investigators' prior pilot study that showed nutrition support improved athlete health and performance metrics. This study has streamlined the protocol and transition to standard-of-care nutrition support to improve scalability and reduce risk to participants.

GENERAL AIMS/HYPOTHESIS: This research program will evidence the importance of nutrition to improve athlete health and performance in Division III athletes. The investigators hypothesize that nutrition screening and support will improve athlete health and performance metrics. As a feasibility study, the primary aim is to assess the feasibility of scaling this nutrition support to a larger student athlete population than the first pilot trial (estimated 100-200 athletes compared to the original 27 from the pilot study). The investigators will assess feasibility from both logistic and financial perspectives. Secondary aims include athlete health and wellness metrics, such as body composition, strength, and health and wellness questionnaires, involving body image, injuries, energy levels and other important mental and physical factors.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: from 18 years of age and up
2. Currently active and NCAA-eligible (including academic standing) member of any Case Western Reserve University (CWRU) Athletic Team
3. Signed Informed Consent

Exclusion Criteria:

1. Under 18 years of age
2. Pregnant women or women who are nursing
3. Unwilling to provide anthropometrics, questionnaires or other collection needs
4. History of a diagnosed disordered eating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | Baseline/Pre-season (August 2025), Mid-season (~2 months after baseline; October 2025), End of Study/End of Competitive Season (~4 months after baseline; December 2025)
  Grip force in kilograms determined by a handgrip dynamometer, conducted on both arms, according to standard practice procedures.

SECONDARY OUTCOMES:
Low Energy Availability in Females Questionnaire (LEAF -Q) | Baseline/Pre-season (August 2025), Mid-season (~2 months after baseline; October 2025), End of Study/End of Competitive Season (~4 months after baseline; December 2025)
  Female participants only. Focuses on physiological symptoms of insufficient energy intake. includes 25 questions arranged in three separate, sequential sections: injuries, gastrointestinal, and reproductive functions. (score; 0-36; total score ≥8 is to be considered at risk)
Low Energy Availability in Males Questionnaire (LEAM -Q) | Baseline/Pre-season (August 2025), Mid-season (~2 months after baseline; October 2025), End of Study/End of Competitive Season (~4 months after baseline; December 2025)
  The low energy availability in males questionnaire (LEAM -Q), focuses on physiological symptoms of relative energy deficiency. Categories include dizziness, gastrointestinal function, thermoregulation at rest, health problems, and recovery. The questionnaire also focuses on physiological symptoms of relative energy deficiency. A higher total score indicates a greater risk of low energy availability. Precise scoring cutoffs are not yet defined.
Body Composition - Fat Mass | Baseline/Pre-season (August 2025), Mid-season (~2 months after baseline; October 2025), End of Study/End of Competitive Season (~4 months after baseline; December 2025)
  Fat mass (kilograms) and as a percent of total body mass.
Body Composition - Fat Free Mass | Baseline/Pre-season (August 2025), Mid-season (~2 months after baseline; October 2025), End of Study/End of Competitive Season (~4 months after baseline; December 2025)
  Fat Free Mass (kilograms) and expressed as a percent of total body mass.
Eating Disorder Examination Questionnaire (EDE-Q) | Baseline/Pre-season (August 2025), Mid-season (~2 months after baseline; October 2025), End of Study/End of Competitive Season (~4 months after baseline; December 2025)
  Measures eating disorder psychopathology. It provides a measure of the range and severity of eating disorder features. (score; continuous beginning at 0; a higher score means greater risk)
Contextual Body Image Questionnaire for Athletes (CBIQA) | Baseline/Pre-season (August 2025), Mid-season (~2 months after baseline; October 2025), End of Study/End of Competitive Season (~4 months after baseline; December 2025)
  Measures four dimensions of body image (Appearance (3 questions), Body Shape (3 questions), Muscularity (3 questions) and Body Weight and Fat (5 questions)) in the context of both athletics and daily life. (7-point Likert scale for each question; scaled scores for each of the four dimensions are obtained by dividing the sum of each question score within that dimension divided by the number of questions in that dimension; scoring is relative to each question with a score of 4 being neutral)
Muscle Dysmorphic Disorder Inventory (MDDI) | Baseline/Pre-season (August 2025), Mid-season (~2 months after baseline; October 2025), End of Study/End of Competitive Season (~4 months after baseline; December 2025)
  The MDDI consists of 13 items addressing drive for size, appearance intolerance, and functional impairment, and serves as a screening tool for muscularity concerns and muscle dysmorphia. Based on a 5-point likert scale. A higher score indicates greater risk for Muscle Dysmorphic Disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Kristyen Tomcik, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request, with appropriate data sharing agreements in place, and according to institutional policy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 12 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
URL: https://case.edu/research/compliance/human-research-protection-program/cwru-institutional-review-board

REFERENCES:
- [Background] Thomas DT, Erdman KA, Burke LM. Position of the Academy of Nutrition and Dietetics, Dietitians of Canada, and the American College of Sports Medicine: Nutrition and Athletic Performance. J Acad Nutr Diet. 2016 Mar;116(3):501-528. doi: 10.1016/j.jand.2015.12.006. PMID 26920240
- [Background] Mountjoy M, Sundgot-Borgen J, Burke L, Carter S, Constantini N, Lebrun C, Meyer N, Sherman R, Steffen K, Budgett R, Ljungqvist A. The IOC consensus statement: beyond the Female Athlete Triad--Relative Energy Deficiency in Sport (RED-S). Br J Sports Med. 2014 Apr;48(7):491-7. doi: 10.1136/bjsports-2014-093502. PMID 24620037